CLINICAL TRIAL: NCT04669327
Title: Hip and Knee Abductor Moments in Normal Subjects and Subjects With Idiopathic Scoliosis: Comparative Study
Brief Title: Hip and Knee Moments Normal and With Scoliosis
Status: Completed | Type: Observational
Sponsor: Taif University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Hatem Allam, Assistant professor, Taif University
Other Study IDs: 331
Record Dates: First submitted 2020-12-05; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Scoliosis Idiopathic
Keywords: Idiopathic scoliosis-gait-moment
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: normal subjects
  Interventions: Other: gait analysis
- Scoliosis: subjects with moderate idiopathic scoliosis
  Interventions: Other: gait analysis

INTERVENTIONS:
Other: gait analysis — Vicon nexus with MTI force plate form

SUMMARY:
Kinetic analysis appears to be useful in providing objective information regarding the gait abilities of scoliotic patients which is difficult to be observed in a clinical setting. Objective: the aim of the study was to analyze the hip and knee peak abductor moments during gait in subjects with idiopathic scoliosis.

DETAILED DESCRIPTION:
The hip and knee abductors' moments normalized to body weight have been investigated in normal subjects and subjects with idiopathic scoliosis. The scoliosis group included a twenty-two-moderate idiopathic dorso-lumbar single scoliotic curve. The control group contained a normal twenty-two subjects. 3D motion analysis system and force plat were used for data collection for hip and knee abductor moment. MANOVA was used to study the difference between normal and scoliotic groups' hip and knee abductor moments in both lower limbs. at alpha level of significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* normal subjects free from any musculoskeletal problems
* subjects with moderate idiopathic scoliosis (cobb angle 25-35)

Exclusion Criteria:

* any musculoskeletal affection rather than scoliosis, neurological manifestations, or previous major surgeries

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: normal subjects and subjects with moderate idiopathic scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
hip and knee abductor moment | one session of 40 minutes.
  peak abductor moment normalized to body weight

CONTACTS AND LOCATIONS:
Overall Officials: HAtem H Allam, Ass. Prof., Principal Investigator — Assistant professor
Locations (1):
- College of Applied Medical Sciences, Ta'if, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
the used consent form indicated that the IPD would be confidential and cannot be published.

REFERENCES:
- [Background] Karol L., Halliday, Gourineni P (2000).: Gait and function after intraarticular hip arthrodesis during a dolescence. J. Bone Joint Surg Am 82: 561-569. Stephen J. and Stricker M. (2002): The Malaligned Adolescent SpinePart 1: Idiopathic Adolescent Scoliosis.International Pediatrics (17): 43-47. Sucato D., Hedequist D. and Karol L(1998).: Gait analysis in idiopathic scoliosis before and after surgery: a comparison of the pre- and postoperative muscle activation pattern. Eur Spine J 7(1): 6-11. Allington N. and Bowen J. (1996): Adolescent idiopathic scoliosis: treatment with the Wilmington brace: A comparison of full-time and part-time use. J Bone Joint Surg 78: 1056-1062. Burwell R., Cole A., Cook T., Grivas T., Kiel A., Moulton A., Thirlwall A., Upadhyay S., Webb J. andWemyss S (2004).: Pathogenesis of idiopathic scoliosis. J Bone Joint Surg 86(9): 2005-2014.